CLINICAL TRIAL: NCT06423261
Title: Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of GB002 Recombinant Polypeptide Inhalation Solution in a Randomized, Double-blind, Placebo-controlled, Dose-increasing Single and Multiple Administration in Chinese Healthy Adult Subjects.
Brief Title: Safety, Tolerability, Pharmacokinetics and Immunogenicity Study of GB002 Recombinant Peptide Inhalation Solution in Healthy Subjects
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Echon Biopharm Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YKSW-GB002-R01
Record Dates: First submitted 2024-04-30; First posted 2024-05-21 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Ascending Dose of GB002 Recombinant Peptide Inhalation Solution (Experimental): Each subject will receive one single administration of GB002 recombinant peptide inhalation solution. The dosage of each group is 0.625mg, 1.25mg, 2.5mg, 5.0mg,7.5mg, respectively.
  Interventions: Drug: GB002 Recombinant Peptide Inhalation Solution; Drug: Placebo
- Multiple Ascending Dose of GB002 Recombinant Peptide Inhalation Solution (Experimental): The subjects will receive multiple doses of GB002 recombinant peptide inhalation solution, administered twice a day for 6 consecutive days. The dosage for each group is 2.5mg, 5.0mg, and 6.5mg, respectively.
  Interventions: Drug: GB002 Recombinant Peptide Inhalation Solution; Drug: Placebo

INTERVENTIONS:
Drug: GB002 Recombinant Peptide Inhalation Solution — Inhalation administration
Drug: Placebo — Inhalation administration

SUMMARY:
This trial is conducted in China. The purpose of this clinical trial is to evaluate the safety and tolerability, pharmacokinetic (PK) characteristics, and immunogenicity of single/multiple inhalation of different doses of GB002 recombinant peptide in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese healthy subjects aged 18 years and above (including 18 years old), both male and female;
2. Male weight ≥50kg, female weight ≥45kg, and body mass index (BMI) in the range of 19-26kg /m² (including the critical value), body mass index (BMI) = weight (kg)/height 2 (m²);
3. Sign informed consent before the test, and fully understand the test content, process and possible adverse reactions;
4. The subjects were able to maintain good communication with the investigators, and understood and complied with the requirements of the clinical trial.

Exclusion Criteria:

1. Participants in any drug clinical trial or use of investigational drug within 3 months prior to the use of investigational drug;
2. Have a history of respiratory disease, such as acute exacerbation of chronic obstructive pulmonary disease, pulmonary fibrosis, pulmonary hypertension, pulmonary hydroedema, pulmonary interstitial disease, bronchial asthma, paradoxical bronchospasm, or throat ulcers, edema, or edema, or have undergone throat, trachea/bronchus, or lung surgery, or within 4 weeks prior to the use of the study drug, Patients with a history of upper and lower respiratory tract infection or acute sinusitis caused by viruses or bacteria, which is considered clinically significant by researchers;
3. Patients with a medical history of cardiovascular system, digestive system, endocrine system, urinary system, nervous system, hematology, immunology (including personal or family history of inherited immune deficiency), metabolic abnormalities, and researchers believe that the current clinical significance;
4. Allergy to any of the ingredients of the drug, or a history of allergy to drugs, foods, pollen or other substances, in particular a known allergy to protein foods, or a history of respiratory allergic disease;
5. Patients who cannot tolerate venipunctures or have a history of fainting needles and fainting blood;
6. Patients who have undergone surgery within 6 months prior to the use of the investigational drug that researchers judge will affect drug absorption, distribution, metabolism, and excretion; Or have undergone surgical procedures within 4 weeks prior to the use of the investigational drug; Or plan to undergo surgical procedures during the study period;
7. Used any drug (including prescription drugs, over-the-counter drugs, Chinese herbs, health care products, etc.) within 14 days before the use of the experimental drug;
8. Persons who have received the vaccine or live attenuated vaccine within 14 days prior to the use of the investigational product, or who plan to receive the vaccine during the trial period;
9. People who donated blood or lost a large amount of blood (>400mL) within 3 months prior to the use of the investigational drug, received blood transfusions or used blood products, or intended to donate blood or blood components during or within 3 months after the end of the trial;
10. Drug abusers or those who have used soft drugs (e.g., cannabis) or hard drugs (e.g., cocaine, PCP, etc.) within one year prior to the use of the investigatory drug;
11. Smokers or smokers who smoked more than 5 cigarettes per day in the 3 months prior to the use of the experimental drug, or who could not stop using any tobacco products during the test period;
12. Alcoholics or regular drinkers in the six months prior to the use of the experimental drug, i.e. drinking more than 14 units of alcohol per week (1 unit =360mL beer or 45mL spirits with 40% alcohol or 150mL wine); Or unwilling to stop drinking alcohol or any products containing alcohol during the trial;
13. Those who consumed excessive amounts of tea, coffee and/or caffeinated beverages (more than 8 cups, 1 cup =250mL) per day, or did not agree to stop drinking tea, coffee and/or caffeinated beverages during the study period;
14. Eat any diet (including grapefruit or grapefruit products, dragon fruit, mango, grapefruit, orange, etc.) that may affect the metabolism of the drug in the body within 7 days prior to the use of the investigatory drug, or any other diet that the researcher considers to affect the absorption, distribution, metabolism or excretion of the drug, or do not agree to stop eating the above diet during the trial period;
15. Those who have special requirements for diet and cannot comply with a unified diet;
16. Subjects (or their partners) have pregnancy plans, sperm and egg donation plans, or do not wish to use one or more non-drug contraceptive methods (such as total abstinence, condoms, pregnancy avoidance rings, partner ligation, etc.) during the trial period to 3 months after the trial ends;
17. Female subjects are pregnant or lactating women; Or had unprotected sex within 2 weeks prior to the use of the investigational drug; Use of oral contraceptives within 30 days prior to the use of the investigational drug or use of long-acting estrogen or progesterone injections or implants within 6 months prior to the use of the investigational drug;
18. Patients with clinically significant abnormalities in physical examination, 12-lead electrocardiogram, vital signs (blood pressure, pulse, body temperature, SpO2), chest X-ray, laboratory examination, and pulmonary function examination (as determined by the clinician);
19. Pulmonary function examination: FEV1 measured value /FEV1 estimated value ≤80% or FVC≤ 80% of the estimated value;
20. Positive results of tobacco test;
21. Positive urine screening test;
22. Positive alcohol breath test;
23. Failure to use the inhalant delivery device correctly or unqualified inhalant delivery training;
24. Subjects may not be able to complete the study for other reasons or may have other reasons deemed inappropriate by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-08-24 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-07-29 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | Day 1 to Day 28

SECONDARY OUTCOMES:
Plasma GB002 Recombinant Peptide concentrations | Day 1 to Day 7
Immunogenicity | Day 14 and Day 28
  Anti-drug antibody（ADA）and neutralizing antibody Nab

OTHER OUTCOMES:
GB002 Recombinant Peptide concentrations in induced sputum | Day 1 to Day 7

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Hospital of Changsha, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No